CLINICAL TRIAL: NCT01208480
Title: A Phase II Trial of Neoadjuvant Bevacizumab, Docetaxel and Carboplatin for Triple Negative Breast Cancer (Neat Trial)
Brief Title: Bevacizumab, Docetaxel, and Carboplatin in Treating Women With Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Joohyuk Sohn, Professor, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000685975; KCSG-0905
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; triple-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Bevacizumab; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Avastin, docetaxel, carboplatin — Avastin, docetaxel, carboplatin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with docetaxel and carboplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with docetaxel and carboplatin works in treating women with operable Stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the rate of pathological complete response in women with operable triple-negative breast cancer treated with neoadjuvant bevacizumab, docetaxel, and carboplatin.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV, docetaxel IV, and carboplatin IV on day 1. Treatment repeat every 3 weeks for 5 courses in the absence of disease progression or unacceptable toxicity. Patients receive docetaxel IV and carboplatin IV only during course 6. Patients undergo surgery between weeks 19-21 as planned.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Stage II or III disease
  * No evidence of metastasis (M0)
  * No inflammatory breast cancer (T4d)
* Must have a primary tumor
* Operable disease
* Triple-negative disease, meeting the following criteria:

  * Estrogen receptor-, progesterone receptor-, and HER2-negative by immunohistochemistry (IHC) 0 or 1+ OR fluorescence in situ hybridization negative (in case IHC is 2+)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Pre- or post-menopausal
* Not pregnant
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥10 g/dL
* Serum creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5 mg/dL
* AST/ALT ≤ 2 times normal
* Alkaline phosphatase ≤ 2 times normal
* Normal or nonspecific EKG
* LVEF ≥ 50% by MUGA or echocardiogram
* Normal mental function to understand and sign the written informed consent
* No history of uncompensated congestive heart failure
* No history of cancer except for carcinoma in situ of the uterine cervix or nonmelanoma skin cancer
* No history or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
* No uncontrolled hypertension (systolic BP > 150 mm Hg and/or diastolic BP > 100 mm Hg)
* No history or evidence of clinically significant cardiovascular disease, including any of the following:

  * Cerebrovascular accident (CVA) or stroke within the past 6 months
  * Myocardial infarction (MI) within the past 6 months
  * Unstable angina
  * NYHA class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
* No serious nonhealing wound, peptic ulcer, or bone fracture
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No known hypersensitivity to any of the study drugs

PRIOR CONCURRENT THERAPY:

* No prior hormone therapy, chemotherapy, or radiotherapy for breast cancer
* No prior breast surgery other than biopsy to confirm diagnosis
* No concurrent chronic daily corticosteroids (more than 10 mg/day methylprednisolone equivalent)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
pathologic complete response (pCR)after completion of 6th cycle neoadjuvant treatment | After completion of 6 cycle of neoadjuvant chemotherapy followed by surgery
  Primary end point in our study is pCR after 6 cycle of neoadjuvant treatment followed by surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joo Hyuk Sohn, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea